CLINICAL TRIAL: NCT04893356
Title: Impact of O6-methylguanine-DNA Methyltransferase (MGMT) Promoter Methylation and MGMT Expression on Dacarbazine Treated Sarcoma Patients (MGMT)
Acronym: MGMT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MGMT
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — O(6)-Methylguanine-DNA Methyltransferase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human DNA will be extracted from tumor tissues using the FFPE DNA Tissue Kit (Qiagen, Hilden, Germany), following the manufacturer's instructions. DNA quality will be checked using NanoDrop 2000 (Thermo Scientific, Waltham, MA, USA). Genomic DNA (500ng) will be converted by sodium bisulfite with the EZ DNA Methylation Gold Kit (Zymo Research, Irvine, CA, USA) and eluted in 20μL RNase free water, according to the manufacturer's instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dacarbazine treated sarcoma patients: Approximately 75 patients with histological diagnosis of Leiomyosarcoma (SCL) and Solitary Fibrous Tumor(SFT), previously treated with dacarbazine alone or associated with anthracyclines, will be enrolled, diagnosed from 2010 to 2020.
  From formalin fixed tumor samples, DNA will be extracted and MGMT expression and MGMT promoter methylation analyzed.
  Interventions: Genetic: O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation and MGMT expression on dacarbazine treated sarcoma patients

INTERVENTIONS:
Genetic: O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation and MGMT expression on dacarbazine treated sarcoma patients — Tumor samples of Leiomyosarcoma and Solitary Fibrous Tumours patients, dacarbazine (as single agents or in combination with anthracyclines) treated, will be obtained from and characterized by the Pathology Unit of the "Istituto Nazionale Tumori Fondazione Pascale" in Naples, Campus Biomedico of Rome, Istituto Oncologico of Bari and University of Palermo.
  Glioblastomas control samples will be obtained from CEINGE-Biotecnologie Avanzate, in Naples and characterized by the Pathology Unit of the University of Naples "Federico II".
  After biopsy or surgical resection, the tissues were fixed in 10% formalin and included in paraffin blocks. All patients partecipating in this study provided informed consent.

SUMMARY:
MGMT study is a retrospective, non-profit, multi-center, observational study. The scientific objective of this study is to investigate whether MGMT expression or MGMT promoter methylation may represent a predictive marker for dacarbazine sensitivity in sarcoma patients.

DETAILED DESCRIPTION:
Sarcomas comprise a group of rare malignancies that are challenging to treat. Incidence of sarcoma is 15,000 annually in the U.S. [1] with a high case fatality rate. Up to one fourth of patients with sarcomas present with metastatic disease, and up to one half of patients who present with locally advanced disease develop metastases despite surgical resection and radiotherapy. Standard chemotherapies (doxorubicin, ifosfamide; gemcitabine and docetaxel) have modest activity with single-agent and combination response rates of 10%-20% and 17%- 40%, respectively .

For patients with primary soft tissue sarcomas, surgery with or without radiotherapy can offer a cure, but nearly half of patients recur and eventually die, with an estimated median survival of 12 to 15 months . As a result, treatment of metastatic or unresectable disease with cytotoxic agents is often given for palliative rather than curative purposes. These cytotoxic agents often incorporate anthracycline- or gemcitabine-based regimens as a first line treatment. Other agents such as dacarbazine and ifosfamide, only show clinical improvement in overall response rate and progression free survival (PFS), without significant benefit in overall survival. Moreover, despite superior PFS observed with these conventional cytotoxic therapies, they are fraught with severe toxicities and attendant high costs, a burden for both patients and health care systems. Until recently, a limited number of drugs have been available for these patients. Doxorubicin and ifosfamide are agents with well established activity that, given sequentially or in combination, constitute the standard treatment of advanced STS. Dacarbazine (DTIC) also is a drug with some classically known activity. The results obtained by using these standard agents, however, remain disappointing, with a median overall survival (OS) close to 12 months.

In the Randomized Phase II Study Comparing Gemcitabine Plus Dacarbazine Versus Dacarbazine Alone in Patients With Previously Treated Soft Tissue Sarcoma, the A Spanish Group for Research on Sarcomas Study showed The combination of gemcitabine and DTIC is active and well tolerated in patients with STS, providing in this phase II randomized trial superior progression-free survival and overall survival than DTIC alone. This regimen constitutes a valuable therapeutic alternative for these patients.

Recent phase III clinical trials have confirmed the efficacy of dacarbazine in the leiomyosarcoma subgroup.

So, despite new drugs such as eribulin, trabectedin, or immunotherapy, dacarbazine remains still one of the most important drugs in the therapeutic landscape of sarcomas, registering in aeterogeneous cases series including liposarcomas and leiomiosarcomas a m PFS 2 ms and a m OS 12 ms , with 10% RR and 60% DCR approximately.

Increased detoxification, activation of general anti-apoptotic pathways, and the activation of repair mechanisms also represent such more general resistance mechanisms to alchylating agents , as dacarbazine and temozolomide. . One of these more general resistance mechanisms is the DNA repair enzyme O6-methylguanine-DNA methyltransferase (MGMT).

MGMT transfers methyl groups from the O6 position of guaninein DNA to a cysteine residue in its active site, thereby inactivating MGMT itself. Inactivated MGMT molecules are ubiquitinatedand degraded by the proteasome. If the methyl group is not removed from guanine, guanine can pair with thymine during DNA replication which leads to transition of guanine-cytosineto adenine-thymine. Cross-linking with cytosine and inhibition ofDNA replication can also occur, leading to apoptotic cell death dueto insufficient DNA repair of point mutations or even chromosomal aberrations and subsequent loss of protein function. Epigenetic changes can also inactivate MGMT by methylationof the associated MGMT gene promoter. Data from clinical trialsfrom patients with glioblastoma demonstrated a strong correlation between methylation of the MGMT promoter and a significantly prolonged survival.

Although this well-established clinical impact of MGMT may also involve radiotherapy and a variety of alkylating agents, the methylation status of the MGMT promoter or MGMT activity is nowadays nearly synonymously used as prognostic predictor for the outcome of glioblastoma patients undergoing chemotherapy withtemozolomide. Temozolomide is animidazotetrazine derivative of dacarbazine. Temozolomide and dacarbazine are both prodrugs that are activated in vivo to the same active compound, monomethyl triazeno imidazole carboxamide (MTIC). MTIC is an alkylating compound that acts mainly by generation of O6-methylguanine. While temozolomide is mainly used for treatment of malignant gliomas and melanomas, darcarbazine represents an effective chemotherapeutic agent for treatment of aggressive and progressive, locally advanced and metastatic sarcomas.

Thus, the primary endpoint of the present project will be to investigate whether MGMT activity or MGMT promoter methylation may also represent a predictive marker for dacarbazine sensitivity of sarcomas .

Retrospectively, will be analysed the expression of MGMT in the present study and the methylation status of the MGMT promoter in hystological sample of 80 patients (LMS and SFT) in correlation with their sensitivity for dacarbazine treatment. In particular, the aim is to demonstrate that MGMT promoter methylation correlates with dacarbazine treatment outcames, studied in terms of response rate and prognosis.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a histological diagnosis of metastatic LMS and SFT from 2010 to 2020, previously treated with dacarbazine alone or with anthracyclines as first line of chemotherapy.

Exclusion Criteria:

* Patients with histological diagnosis of metastatic LMS and SFT, received before 2010.
* Patients with histological diagnosis of metastatic LMS and SFT from 2010 to 2020, never treated with dacarbazine
* Patients with a histological diagnosis of metastatic LMS and SFT from 2010 to 2020, previously treated with dacarbazine alone or with anthracyclines as the first line of chemotherapy, of which, however, there is no tissue sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor specimens from patients with Leiomyosarcoma (SCL) and Solitary Fibrous Tumors (SFT), treated with dacarbazine (as a single agent or in combination with anthracyclines), after biopsy or surgical resection, are fixed in 10% formalin and included in blocks of paraffin. They will be compared with control samples of glioblastomas (provided by the CEINGE-Biotechnologies Advanced, of Naples).
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
To analyze the expression of the MGMT gene in patients with Leiomyosarcoma (AML) and with metastatic Solitary Fibrous Tumor (SFT) | 1 year
To analyze the methylation status of the MGMT promoter in histological specimens | 1 year

SECONDARY OUTCOMES:
To investigate whether MGMT activity or MGMT promoter methylation may also represent a predictive marker for dacarbazine sensitivity in sarcomas | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute of Naples, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No